CLINICAL TRIAL: NCT03457558
Title: Assessment of Food Security and Perceptions and Barriers to Healthy Eating in Individuals With Spinal Cord Injuries Living in the Community
Brief Title: Food Security and Perceptions and Barriers to Healthy Eating in Individuals With Spinal Cord Injuries
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 05-17-21E
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Food security is one's ability to get food. Individuals with a Spinal Cord Injury (SCI) have many risk factors for low rates of food security. Some of these risk factors include lower levels of income and employment. Our long-term goal is to identify if food security is more prevalent in the SCI population, and to develop ways to improve food security in the SCI population. The purpose of this study is to determine the rates of food insecurity in a sample of people living with a SCI and to identify some perceptions of barriers to healthy eating in the SCI population.

DETAILED DESCRIPTION:
Food security is one's ability to get food. Individuals with a SCI have many risk factors for low rates of food security. Some of these risk factors include lower levels of income and employment. This study consists of a one-time survey using the US Adult Food Security Survey and another previously validated survey about perceptions of barriers to healthy eating.

Our long-term goal is to develop a large SCI food security and perceived barriers to healthy eating multicenter study in order to determine if these factors are significant issues in the SCI population. We also aim to determine the causes of these issues in order to develop interventions to improve the health of all people living with a SCI and potentially reduce their health care costs. The purpose of this study is to determine the rates of food insecurity in a sample of people living with a SCI and to identify some perceptions of barriers to healthy eating in the SCI population. This will also develop preliminary data to support a NIH R level grant application for a large, multicenter study to further explore SCI food security at the national level. Our central hypothesis is that there will be an increased rate of food insecurity in the SCI population compared to other groups in the literature, and that this will be associated with income and environmental barriers.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* Male or female, any ethnicity, with the history of a spinal cord injury at least one year prior (without a diagnosis of Multiple Sclerosis or malignant cancer)
* Community wheelchair user
* Voluntary, informed consent of participant and interest in participating in further research studies
* Lives in the community, not a skilled nursing facility

Exclusion Criteria:

* age <18 years old
* Chronic, nontobacco substance-abuse
* Community ambulator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults, >18 years of age, of any ethnicity and race, with history of a SCI without the diagnosis of multiple sclerosis or malignant cancer, at least one year prior to enrollment in the study. All participants will be community wheelchair users.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Food Security | Completed at time of enrollment
  The US Adult Food Security Survey will be administered to all participants. They will each receive a score of 0-10. A score of zero represents high food security. A score of 1-2 represents marginal food security. A score of 3-5 represents low food security, and a score of 6-10 represents very low food security.
Perception Barriers | Completed at time of enrollment
  Perceived personal, social, and environmental barriers will be measured using a questionnaire previously used among young women

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Lieberman, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Rehabilitation, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No